CLINICAL TRIAL: NCT04918628
Title: A Safety and Efficacy Study of Neoadjuvant Chemotherapy Combined With CCRT Followed by Adjuvant Chemotherapy and Anti-PD-1 Antibody in Patients With Stage IIIC2-IVB Cervical Cancer
Brief Title: Adjuvant Chemotherapy and Anti-PD-1 Antibody in Patients With Stage IIIC2-IVB Cervical Cancer
Acronym: CRTCP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Head of Department of Radiation Oncology, Chief Physician, Taizhou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHH-202105
Record Dates: First submitted 2021-05-28; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Neoadjuvant Chemotherapy Combined With CCRT Followed by Adjuvant Chemotherapy and Anti-PD-1 Antibody(Sintilimab 200mg intravenous drip every three weeks until PD or 2 years).
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — A humanized anti-PD-1 monoclonal antibody

SUMMARY:
This phase II study is to Evaluate the Safety and Efficacy of Neoadjuvant Chemotherapy Combined With CCRT Followed by Adjuvant Chemotherapy and Anti-PD-1 Antibody in Patients With Stage IIIC2-IVB Cervical Cancer.（ CRTCP）

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of adjuvant chemotherapy and anti-PD-1 antibody combined with CCRT in patients with stage IIIC2-IVB cervical cancer.

SECONDARY OBJECTIVES:

I. To investigate the feasibility of administration of chemotherapy and anti-PD-1 antibody as a adjuvant therapy with chemoradiation (CRT) therapy in patients with stage IIIC2-IVB cervical cancer.

II. To determine the nature and degree of toxicity of chemotherapy and anti-PD-1 antibody as a adjuvant therapy with chemoradiation (CRT) therapy in patients with stage IIIC2-IVB cervical cancer.

III. To examine the changes in T cell receptor (TCR) clonality, diversity, and frequency in peripheral blood and tissue and correlate this with clinical outcomes, such as the exploratory response assessment on the post-treatment positron emission tomography (PET)-computed tomography (CT) scan and 2-year Progression-Free Survival (PFS).

IV. To assess the predictive value of baseline and on-treatment PD-L1 expression in the tissue in each treatment arm for clinical outcomes using post-treatment PET-CT scan and 2-year PFS as the outcome measures.

EXPLORATORY OBJECTIVES:

I. To explore baseline and on-treatment blood and tissue biomarkers that could predict response to the combination therapy and 2-year PFS.

II. To explore the response assessment on the exploratory and the clinical 2-year Progression-Free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to any protocol-related procedures.
2. Aged 18-75 years(including 18 years old and 75 years old).
3. Bodyweight of greater than 30 kg.
4. Must have an average life expectancy of 6 months.
5. Histologically or cytologically confirmed advanced/metastatic cervical cancer.
6. Eastern Cooperative Oncology Group (ECOG) ≤ 2 or Karnofsky Performance Status of ≥ 60.
7. Participants must have normal organ and marrow function as defined below: (Hgb >=9g/dl, Absolute neutrophil count ≥1500/mcL, Platelets ≥100000/mcL, Total bilirubin <=1.5 x normal institutional limits, AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal, Creatinine clearance >40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976).

   -

Exclusion Criteria:

1. Female patients who are pregnant or breastfeeding or female patients of reproductive potential who are not willing to employ effective birth control.
2. History of prior malignancy within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as but not limited to, non-melanoma skin carcinoma, ductal carcinoma in situ, or stage I endometrioid uterine cancer, and others at the discretion of the Principal Investigator (PI).
3. Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases are permissible. Patients with untreated brain metastases, spinal cord compression, or leptomeningeal carcinomatosis are excluded from this clinical trial because of their poor prognosis, because of symptoms that may arise from inflammatory reactions, and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with brain metastases or spinal cord compression previously treated with radiation and/or surgery are allowed if local treatment was >30 days ago, most recent MRI demonstrates stability or decrease in size of all lesions, and the patient has no current neurologic symptoms related to the metastases and treatment and no requirement for corticosteroids related to the prior treatment.
4. Prior oncology vaccine therapy.
5. History of allogeneic organ transplantation.
6. Subject has an immunodeficiency.

(1) Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF)-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of the need for systemic immunosuppressive medication during the course of the study, with the following exceptions: Patients who received acute, low-dose systemic immunosuppressant medication（exceed 10 mg/day of prednisone or its equivalent） or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency.

(2)Subject has an active autoimmune disease in the past 2 years. (3)Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroid disease, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions: Patients with a history of autoimmune-related hypothyroidism who are on the thyroid replacement hormone are eligible for the study; Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

7.Treatment with a vascular endothelial growth factor (VEGF) inhibitor within the last 6 weeks.

8.Major surgical procedure (as defined by the treating physician) within 28 days prior to the first dose of ICIs or still recovering from prior surgery.

9.Active or prior documented interstitial lung disease.

10.History of hypersensitivity to ICIs or any CTLA4, PD1, or PDL-1 inhibitor.

11.Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies); patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible; patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).

12.History of prior bowel fistula, ulcerations, or perforations. 13.Any medical, psychological, or social condition that in the opinion of the treating physician would interfere with the evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Grade 3 and Grade 4 Treatment-related adverse events (TRAEs) | From screening till final visit (upto a maximum of 24 months)
  To assess the safety and tolerability profile of Sintilimab as defined by Grade 3 and Grade 4 TRAEs within 6 months from the initiation of durvalumab Sintilimab treatment

SECONDARY OUTCOMES:
Median Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by the Investigator | From the first date of treatment until the date of objective disease progression or death (up to maximum 24 months)
  To assess the efficacy of Sintilimab treatment in terms of PFS. PFS will be calculated using Kaplan-Meier product limit methods.
PFS at 24 months (PFS24) | From the first date of treatment until the date of objective disease progression or death (up to maximum 24 months)
  To assess the efficacy of Sintilimab treatment in terms of PFS. PFS will be calculated using Kaplan-Meier product limit methods.
Median overall survival (OS) | From the first date of treatment until death due to any cause (up to maximum 24 months)
  To assess the efficacy of Sintilimab treatment in terms of OS. OS will be calculated using Kaplan-Meier product limit methods.
OS at 24 months (OS24) | Time Frame: From the first date of treatment until death due to any cause (up to maximum 24 months)
  To assess the efficacy of Sintilimab treatment in terms of OS. OS will be calculated using Kaplan-Meier product limit methods.
Number of participants with immunological colitis | From screening till final visit (up to a maximum of 24 months)
  To assess the safety and tolerability profile of Sintilimab treatment in terms of the number of participants with abnormal immunological colitis. Immunological colitis will be collected before, during, and after Sintilimab infusion. Fecal occult blood test to assess gastrointestinal bleeding, gastrointestinal angiography to assess gastrointestinal perforation.
Number of participants with immunological rash | From screening till final visit (up to a maximum of 24 months)
  To assess the safety and tolerability profile of Sintilimab treatment in terms of the number of participants with abnormal immunological rash. Immunological rash will be collected before, during, and after Sintilimab infusion.
Number of participants with abnormal blood pressure (BP) | From screening till final visit (up to a maximum of 24 months)
  To assess the safety and tolerability profile of Sintilimab treatment in terms of the number of participants with abnormal BP. BP will be collected before, during, and after IP infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Sufang Wu, MD, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Locations (1):
- Youyou Xie, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No